CLINICAL TRIAL: NCT05997108
Title: Platelet and Red Blood Cell Volume Indices as Inflammatory Biomarkers in Ankylosing Spodylitis
Brief Title: Platelet and Red Blood Cell Volume Indices as Inflammatory Biomarkers in Ankylosing Spondylitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Margo Gerges Mofeed, Resident-rheumatology department-sohag general hospital, Sohag University
Other Study IDs: Soh-Med-23-07-01MS
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases group
  Interventions: Diagnostic Test: CBC
- control group
  Interventions: Diagnostic Test: CBC

INTERVENTIONS:
Diagnostic Test: CBC — Platelet and red blood cell volume indices

SUMMARY:
this study aims to determine the relatioships among the NLR ,PLR ,MLR ,red cell volume and platelet volume indices levels as biomarkers in ankylosing spondylitis.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT WITH DISEASE DURATION OF MORE THAN 6 MONTHS
* AGE MORE THAN 18 YEARS

Exclusion Criteria:

* PATIENT WITH CARDIAC ,CEREBROVASCULAR AND HEMATOLOGIC DIEASE
* PTIENT WITH HYPERTENSION ,DIABETES ,METABOLIS SYNDROMES AND OTHER AUTOIMMUNE RHEUMATIC DISEASES.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PATIENT WITH DISEASE DURATION OF MORE THAN 6 MONTHS
  -AGE MORE THAN 18 YEARS
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
platelet | 6 months
  platelet cell volume indices
Red blood cell | 6 months
  red blood cell volume indices

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

REFERENCES:
- [Background] Azab B, Torbey E, Singh J, Akerman M, Khoueiry G, McGinn JT, Widmann WD, Lafferty J. Mean platelet volume/platelet count ratio as a predictor of long-term mortality after non-ST-elevation myocardial infarction. Platelets. 2011;22(8):557-66. doi: 10.3109/09537104.2011.584086. Epub 2011 Jun 30. PMID 21714700
- [Background] Coutant F, Miossec P. Evolving concepts of the pathogenesis of rheumatoid arthritis with focus on the early and late stages. Curr Opin Rheumatol. 2020 Jan;32(1):57-63. doi: 10.1097/BOR.0000000000000664. PMID 31644463
- [Background] Bekdas M, Goksugur SB, Sarac EG, Erkocoglu M, Demircioglu F. Neutrophil/lymphocyte and C-reactive protein/mean platelet volume ratios in differentiating between viral and bacterial pneumonias and diagnosing early complications in children. Saudi Med J. 2014 May;35(5):442-7. PMID 24825803
- [Background] Kumano Y, Hasegawa Y, Kawahara T, Yasui M, Miyoshi Y, Matsubara N, Uemura H. Pretreatment Neutrophil to Lymphocyte Ratio (NLR) Predicts Prognosis for Castration Resistant Prostate Cancer Patients Underwent Enzalutamide. Biomed Res Int. 2019 Jan 20;2019:9450838. doi: 10.1155/2019/9450838. eCollection 2019. PMID 30800682